CLINICAL TRIAL: NCT03263429
Title: Phase I/II Study to Evaluate the Safety, Efficacy, and Novel PET/CT Imaging Biomarkers of CB-839 in Combination With Panitumumab and Irinotecan in Patients With Metastatic and Refractory RAS Wildtype Colorectal Cancer
Brief Title: Novel PET/CT Imaging Biomarkers of CB-839 in Combination With Panitumumab and Irinotecan in Patients With Metastatic and Refractory RAS Wildtype Colorectal Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Calithera Biosciences, Inc (Industry)
Responsible Party: Principal Investigator, Jordan Berlin, MD, Principal Investigator, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICC GI 1703; NCI-2017-01461 (Registry Identifier: NCI, Clinical Trials Reporting Program)
Record Dates: First submitted 2017-08-23; First posted 2017-08-28 (Actual); Results first posted 2024-08-30 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Colorectal Cancer; Metastatic Colorectal Cancer; RAS Wild Type Colorectal Cancer; Refractory Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — CB-839; Panitumumab; Irinotecan; Diagnostic Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Panitumumab/Irinotecan/CB-839 (Experimental): Patients receive glutaminase inhibitor CB-839 PO BID on days 1-28, panitumumab IV over 60-90 minutes on days 1 and 15, and irinotecan hydrochloride IV over 90 minutes on day 1 and 15 (Phase I only). Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Glutaminase Inhibitor CB-839; Biological: Panitumumab; Drug: Irinotecan Hydrochloride (phase I only); Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Device: Imaging with 11C-Glutamine PET/CT scans and 18F-FSPG PET/CT scans

INTERVENTIONS:
Drug: Glutaminase Inhibitor CB-839 — Given by mouth
Biological: Panitumumab — Given by vein
Drug: Irinotecan Hydrochloride (phase I only) — Given by vein
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Device: Imaging with 11C-Glutamine PET/CT scans and 18F-FSPG PET/CT scans — During phase II at baseline and day 28 of cycle 1

SUMMARY:
This phase I/II trial studies the best dose and side effects of glutaminase inhibitor CB-839 and how well it works with panitumumab and irinotecan hydrochloride (phase I only) in treating patients with RAS wildtype colorectal cancer that has spread to other places in the body and does not respond to treatment. Glutaminase inhibitor CB-839 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as panitumumab, may interfere with the ability of tumor cells to grow and spread. Drugs used in chemotherapy, such as irinotecan hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving glutaminase inhibitor CB-839 with panitumumab and irinotecan hydrochloride may work better in treating patients with colorectal cancer.

DETAILED DESCRIPTION:
Objectives:

Primary Objective of Phase I:

• Determine the safety and tolerability of CB-839 in combination with panitumumab and irinotecan.

Exploratory Objective of Phase I (Optional Imaging Sub-study):

• Correlate radiological features of pre- and post-treatment 11C-Glutamine PET/CT and 18F-FSPG PET/CT with clinical outcome.

Primary Objective of Phase II:

• Determine the efficacy of CB-839 in combination with panitumumab as measured by the response rate (RR).

Secondary Objectives of Phase II:

* Determine the disease control rate (DCR), progression-free survival (PFS), and overall survival (OS).
* Perform the following correlative studies (in the phase 2 component):
* Correlate radiological features of pre- and post-treatment 18F-FSPG PET/CT with clinical outcome and biological correlates (tissue gene signature, exosomes).
* Collect blood samples during each radiotracer injection to assess pharmacokinetics.
* Collect pre-treatment biopsy tissue and prospectively correlate clinical outcome with a glutamine metabolism gene signature.
* Quantify exosomal content in the plasma.

Exploratory Objective of Phase II:

• Development of patient-derived organoids from pre-treatment tissue biopsy

OUTLINE: Phase I is a dose-escalation study of glutaminase inhibitor CB-839 in combination with standard doses of panitumumab and irinotecan hydrochloride. Phase II will study efficacy of glutaminase inhibitor CB-839 in combination with standard doses of panitumumab.

Patients receive glutaminase inhibitor CB-839 orally (PO) twice daily (BID) on days 1-28, panitumumab intravenously (IV) over 60-90 minutes on days 1 and 15, and irinotecan hydrochloride IV over 90 minutes on day 1 and 15 (Phase I only). Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed at 28 days and then every 3 months for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated written informed consent
* Histologically or cytologically-confirmed diagnosis of metastatic KRAS wildtype colorectal cancer (CRC)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* In dose escalation, patients must have had at least one prior line of chemotherapy for advanced disease or progressed within 6 months of adjuvant therapy (prior chemotherapy and/or anti-EGFR therapy is permitted)
* In dose expansion, patients must have received prior anti-EGFR therapy and achieved at least stable disease on at least one scan as their best response
* In dose expansion, patients must be willing to undergo a pre-treatment biopsy, and four research PET imaging techniques (11C-Glutamine and 18F-FSPG), two pre-treatment and two after one cycle of treatment
* In dose expansion, at least one measurable lesion as defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 which can be followed by CT or magnetic resonance imaging (MRI)
* Absolute neutrophil count (ANC) >= 1,500/uL
* Platelets >= 100,000/uL
* Serum albumin >= 3.0 g/dL
* Serum creatinine =< 2 mg/dL, or calculated creatinine clearance > 50 mL/min (per the Cockcroft-Gault formula)
* Total bilirubin =< 1.5 times upper limit of normal (ULN)
* Aspartate transaminase (AST) and alanine aminotransferase (ALT) =< 5.0 x ULN
* Women of childbearing potential (WOCBP) must have a negative serum pregnancy test within 14 days prior to receiving first dose of protocol-indicated treatment; and additionally agree to use at least 2 methods of acceptable contraception or abstain from heterosexual intercourse from the time of signing consent, and until 2 months after patient's last dose of protocol-indicated treatment; WOCBP of childbearing potential are defined as those not surgically sterile or not post-menopausal (i.e. if a female patient has not had a bilateral tubal ligation, a bilateral oophorectomy, or a complete hysterectomy; or has not been amenorrheic for 12 months in the absence of an alternative medical cause, then patient will be considered a female of childbearing potential); postmenopausal status in females under 55 years of age should be confirmed with a serum follicle-stimulating hormone (FSH) level within laboratory reference range for postmenopausal women
* Men able to father children who are sexually active with WOCBP must agree to use at least 2 methods of acceptable contraception from the time of signing consent and until 2 months after patient's last dose of protocol-indicated treatment; men able to father children are defined as those who are not surgically sterile (i.e. patient has not had a vasectomy)

Exclusion Criteria:

* Within 28 days before first dose of protocol-indicated treatment:

  * Anti-cancer treatment including chemotherapy, radiation, hormonal therapy, targeted therapy, immunotherapy, or biological therapy
  * Major surgery requiring general anesthesia; (Note: within this time frame, placement of a central line or portacath is acceptable and does not exclude)
  * Receipt of an investigational agent
* Within 14 days before first dose of protocol-indicated treatment:

  * Active uncontrolled infection; patients with infection under active treatment and controlled with antibiotics initiated at least 14 days prior to initiation of protocol-indicated treatment are not excluded (e.g. urinary tract infection controlled with antibiotics)
* Dose escalation only: known grade 4 toxicity probably or definitely attributed to past irinotecan treatment
* Active inflammatory bowel disease, other bowel disease causing chronic diarrhea (defined as > 4 loose stools per day), or bowel obstruction
* History of interstitial pneumonitis or pulmonary fibrosis, or evidence of interstitial pneumonitis or pulmonary fibrosis on baseline chest CT scan
* Unable to receive oral medication
* Central nervous system (CNS) metastasis, unless asymptomatic or previously treated and stable; and no evidence of CNS progression for at least 30 days prior to initiating protocol-indicated treatment; anticonvulsant and/or corticosteroid therapy will be allowed if patient is on a stable or decreasing dose of such treatment for at least 30 days prior to initiating protocol-indicated treatment
* Patients with known Gilbert's disease
* Patient is pregnant or breastfeeding
* Current or previous malignant disease (other than colorectal cancer) within the last 5 years; with the exception of the following if considered curatively treated: non-melanoma skin cancer(s), carcinoma in situ of the cervix, and ductal carcinoma in situ; subjects with another active malignancy requiring concurrent anti-cancer intervention are excluded; (Note the following does not exclude: effectively treated malignancy that has been in remission for more than 5 years and is considered to be cured AND no additional anti-cancer therapy is ongoing and required during the study period)
* Known positive test for human immunodeficiency virus (HIV), acquired immunodeficiency syndrome (AIDS), hepatitis A, hepatitis B, hepatitis C, or cytomegalovirus (CMV)
* Known psychiatric condition, social circumstance, or other medical condition reasonably judged by the patient's study physician to unacceptably increase the risk of study participation; or to prohibit the understanding or rendering of informed consent or anticipated compliance with scheduled visits, treatment schedule, laboratory tests and other study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2017-08-23 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Berlin, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (1):
- Vanderbilt-Ingram Cancer Center, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- CB-839 600mg +Panitumumab 6mg/kg +Irinotecan 180mg/m2 (Phase I Dose Escalation): Participants who were treated with CB-839 600mg +Panitumumab 6mg/kg +Irinotecan 180mg/m2
- CB-839 800mg +Panitumumab 6mg/kg +Irinotecan 180mg/m2 (Phase I Dose Escalation); CB-839 800mg +Panitumumab 6mg/kg +Irinotecan180mg/m2 (Phase II Dose Expansion): Participants were treated with CB-839 800mg +Panitumumab 6mg/kg +Irinotecan 180mg/m2
Period: Overall Study
Arm/Group | CB-839 600mg +Panitumumab 6mg/kg +Irinotecan 180mg/m2 (Phase I Dose Escalation) | CB-839 800mg +Panitumumab 6mg/kg +Irinotecan 180mg/m2 (Phase I Dose Escalation) | CB-839 800mg +Panitumumab 6mg/kg +Irinotecan180mg/m2 (Phase II Dose Expansion)
Started | 3 | 8 | 18
Completed | 0 | 0 | 0
Not Completed | 3 | 8 | 18
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Follow-Up Period Completed | 0 | 2 | 0
Not completed — Death | 3 | 5 | 16
Not completed — Participant unable to return | 0 | 0 | 1
Not completed — Study Closed | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CB-839 600mg +Panitumumab 6mg/kg +Irinotecan 180mg/m2 (Phase I Dose Escalation) | CB-839 800mg +Panitumumab 6mg/kg +Irinotecan 180mg/m2 (Phase I Dose Escalation) | CB-839 800mg +Panitumumab 6mg/kg +Irinotecan180mg/m2 (Phase II Dose Expansion) | Total
Number analyzed (Participants) | 3 | 8 | 18 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 16 | 19
  >=65 years | 1 | 7 | 2 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5 | 10
  Male | 2 | 4 | 13 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 1 | 4
  White | 2 | 5 | 13 | 20
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 4 | 4
Region of Enrollment [Number; unit: participants]
  United States | 3 | 8 | 18 | 29

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (Phase I) of CB-839 in Combination With Panitumumab and Irinotecan Hydrochloride
Description: The maximum tolerated dose of CB-839 will be determined in Phase I with dose-escalation following Bayesian continual reassessment method. Patients were treated in cohort of 3. The CB839 dose leves were 400, 600 and 800mg.
Time Frame: Up to 12 months
Population: Patients got CB-839 combined with 6 mg/kg panitumumab, and 180 mg/m2 irinotecan.
Measure: Number; unit: mg
Arm/Group | Panitumumab/Irinotecan/CB-839
Number analyzed (Participants) | 11
mg | 800

2. Primary Outcome: Response Rate (Phase II)
Description: The percent of patients with best response as complete response (CR) and partial response(PR) among patients with evaluable result. The response criteria: CR, Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm; PR, At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters, Progressive Disease (PD), At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition, the sum must also demonstrate an absolute increase of at least 5 mm. (The appearance of one or more new lesions is also considered progression); Stable Disease(SD), Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Time Frame: Up to 12 months
Population: Participants were treated with CB-839 800mg +Panitumumab 6mg/kg +Irinotecan 180mg/m2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CB-839 800mg +Panitumumab 6mg/kg +Irinotecan180mg/m2 (Phase II Dose Expansion)
Number analyzed (Participants) | 17
percentage of participants | 11.8 [3.3 to 34.3]

3. Primary Outcome: Recommended Phase 2 Dose of CB-839 in Combination With Panitumumab and Irinotecan Hydrochloride (Phase I)
Description: The recommended phase 2 dose will be determined.
Time Frame: Up to 12 months.
Population: Patient received CB-839 in combination with panitumumab and irinotecan hydrochloride (Phase I)
Measure: Number; unit: mg
Arm/Group | Panitumumab/Irinotecan/CB-839
Number analyzed (Participants) | 11
mg | 800

4. Secondary Outcome: Disease Control Rate
Description: The disease control rate will be evaluated. It is defined as the percent of patients with response as CR, PR, or SD among patients with evaluable result. The response criteria: CR, Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm; PR, At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters, Progressive Disease (PD), At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition, the sum must also demonstrate an absolute increase of at least 5 mm. (The appearance of one or more new lesions is also considered progression); Stable Disease(SD), Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Time Frame: Up to 12 months
Population: Participants were treated with CB-839 800mg +Panitumumab 6mg/kg +Irinotecan 180mg/m2.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CB-839 800mg +Panitumumab 6mg/kg +Irinotecan180mg/m2 (Phase II Dose Expansion)
Number analyzed (Participants) | 17
percentage of participants | 41.2 [21.6 to 64.0]

5. Secondary Outcome: Coefficient of Determination (R2) of Maximum Standardized Uptake Value (SUVmax) of Fluorine F 18 L-glutamate Derivative BAY94-9392 (18F-FSPG) Uptake Change With Tumor Size Change (Phase II)
Description: Evaluate the relationship between 18F-FSPG uptake change from baseline and change in tumor size at the time of objective response assessment using a standard linear regression analysis. The coefficient of determination (R2) describes the strength of the relationship between the change in 18F-FSPG and the change in tumor size. The squared root of R2 is the correation coefficient between the change in 18F-FSPG and the change in tumor size. R2 is reported.
Time Frame: Up to 8 weeks
Population: Patients received the phase II dose and had both SUVmax and tumor size data available
Measure: Number; unit: Coefficient of determination
Arm/Group | CB-839 800mg +Panitumumab 6mg/kg +Irinotecan180mg/m2 (Phase II Dose Expansion)
Number analyzed (Participants) | 7
Coefficient of determination | 0.0983

6. Secondary Outcome: Plasma Exosomal Content (Phase II)
Description: Plasma exosomal content will be assessed at pre-treatment, after one cycle of treatment, and at disease progression.
Time Frame: Up to 12 months
Population: Patients who were treated with CB-839 800mg +Panitumumab 6mg/kg +Irinotecan180mg/m2 and had plasma exosomal measurement available at pre-treatment, after cycle 1, and/or at progression.
Measure: Mean (95% Confidence Interval); unit: mg
Groups:
- CB-839 800mg +Panitumumab 6mg/kg +Irinotecan180mg/m2 (Phase II Dose Expansion) Pre-treatment: Participants were treated with CB-839 800mg +Panitumumab 6mg/kg +Irinotecan 180mg/m2, and had plasma exosomal measurement available at pre-treatment
- CB-839 800mg +Panitumumab 6mg/kg +Irinotecan180mg/m2 (Phase II Dose Expansion) After Cycle 1: Participants were treated with CB-839 800mg +Panitumumab 6mg/kg +Irinotecan 180mg/m2 (Phase II Dose Expansion) and had plasma exosomal content measurement available after cycle 1
- CB-839 800mg +Panitumumab 6mg/kg +Irinotecan180mg/m2 (Phase II Dose Expansion) at Progression: Participants were treated with CB-839 800mg +Panitumumab 6mg/kg +Irinotecan 180mg/m2 (Phase II Dose Expansion) and had plasma exosomal content measurement available at progression
Arm/Group | CB-839 800mg +Panitumumab 6mg/kg +Irinotecan180mg/m2 (Phase II Dose Expansion) Pre-treatment | CB-839 800mg +Panitumumab 6mg/kg +Irinotecan180mg/m2 (Phase II Dose Expansion) After Cycle 1 | CB-839 800mg +Panitumumab 6mg/kg +Irinotecan180mg/m2 (Phase II Dose Expansion) at Progression
Number analyzed (Participants) | 17 | 9 | 7
mg | 3.9 [3.5 to 4.4] | 3.2 [2.7 to 3.7] | 4.1 [3.6 to 4.5]

7. Secondary Outcome: Progression Free Survival (Phase II)
Description: It is defined as the time from on treatment to disease progression or death (whichever comes first). For those alive without progression, they were censored at last follow up date. Kaplan-Meier method was used to estimate the median survival time with 95% confidence interval.
Time Frame: Up to 12 months
Population: Patients received CB-839 800mg +Panitumumab 6mg/kg +Irinotecan180mg/m2.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | CB-839 800mg +Panitumumab 6mg/kg +Irinotecan180mg/m2 (Phase II Dose Expansion)
Number analyzed (Participants) | 17
days | 56 [43 to 93]

8. Secondary Outcome: Overall Survival
Description: It is defined as the days from on treatment date to death due to any cause. Those alive were censored at the last date of follow up. Kaplan-Meier method was used to estimate the median survival time with 95% confidence interval.
Time Frame: Up to 12 months
Population: Patients received CB-839 800mg +Panitumumab 6mg/kg +Irinotecan180mg/m2
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | CB-839 800mg +Panitumumab 6mg/kg +Irinotecan180mg/m2 (Phase II Dose Expansion)
Number analyzed (Participants) | 17
days | 265 [113 to 399]

ADVERSE EVENTS:
Time Frame: Adverse events collected from initiation of protocol-indicated treatment through 28 days after the last dose of protocol-indicated treatment up to approximately 60 months.
Arm/Group | CB-839 600mg +Panitumumab 6mg/kg +Irinotecan 180mg/m2 (Phase I Dose Escalation) | CB-839 800mg +Panitumumab 6mg/kg +Irinotecan 180mg/m2 (Phase I Dose Escalation) | CB-839 800mg +Panitumumab 6mg/kg +Irinotecan180mg/m2 (Phase II Dose Expansion)
All-Cause Mortality (participants affected / at risk) | 3/3 | 8/8 | 17/18
Serious Adverse Events (participants affected / at risk) | 1/3 | 3/8 | 4/18
Other Adverse Events (participants affected / at risk) | 3/3 | 8/8 | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CB-839 600mg +Panitumumab 6mg/kg +Irinotecan 180mg/m2 (Phase I Dose Escalation) (N=3) | CB-839 800mg +Panitumumab 6mg/kg +Irinotecan 180mg/m2 (Phase I Dose Escalation) (N=8) | CB-839 800mg +Panitumumab 6mg/kg +Irinotecan180mg/m2 (Phase II Dose Expansion) (N=18)
Bowel obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Neutrophil Count Decrease (Investigations) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Kidney Injury (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Difficile: related to antibiotic use (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Biliary Obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Brain Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Venting G Tube Complication (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Spouse pregnant (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CB-839 600mg +Panitumumab 6mg/kg +Irinotecan 180mg/m2 (Phase I Dose Escalation) (N=3) | CB-839 800mg +Panitumumab 6mg/kg +Irinotecan 180mg/m2 (Phase I Dose Escalation) (N=8) | CB-839 800mg +Panitumumab 6mg/kg +Irinotecan180mg/m2 (Phase II Dose Expansion) (N=18)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 3 (3) | 3 (4)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 3 (4) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 6 (6) | 2 (2)
Alanine aminotransferase increased (Investigations) | 2 (3) | 3 (5) | 7 (14)
Alkaline phosphtase increased (Investigations) | 2 (3) | 5 (8) | 7 (7)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 3 (6) | 7 (17) | 8 (21)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 3 (4) | 4 (5)
Anxiety (Psychiatric disorders) | 1 (1) | 3 (3) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 3 (7) | 7 (12)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 2 (3)
Bladder spasm (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 1 (1) | 3 (3)
Blurry vision (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Body aches (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Chills (General disorders) | 1 (1) | 2 (2) | 0 (0)
Colonic fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Colonic obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 5 (6) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1)
Cracking of nail and tips of fingers (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Cracks on heels (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 3 (6) | 1 (2)
Cuticle and nail irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 2 (3)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Diabetes (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 6 (10) | 5 (6)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1)
Dry eye (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (2) | 3 (3)
Dysgeusia (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 5 (8)
Limb edema (General disorders) | 1 (2) | 3 (3) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Right eye ulcer (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eyelid irritation (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 3 (4) | 7 (10) | 9 (19)
Facial pain (General disorders) | 0 (0) | 2 (2) | 0 (0)
Fever (General disorders) | 1 (1) | 2 (2) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 4 (4) | 0 (0)
Cracking on feet (General disorders) | 1 (1) | 0 (0) | 0 (0)
Groin muscle pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Hand fissure (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 3 (3) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (4) | 8 (11) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 13 (22)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 2 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 4 (7) | 3 (9)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 3 (6) | 5 (9) | 7 (11)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 3 (5) | 7 (9)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 3 (5) | 2 (3)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 3 (4) | 0 (0)
Left femur pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (2) | 5 (12) | 7 (11)
Memory impairment (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 2 (2) | 4 (4) | 1 (1)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal conjestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 5 (5) | 9 (9)
Neck edema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (2) | 4 (8) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Palpatations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2)
Stab wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Eye lash growth (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Abdominal Cramping (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Possible bleeding in the GI tract (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Discomfort to light exposure (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Welts on ankle and calf (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin is splitting on hands and feet (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Seborrheic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 1 (1) | 3 (4) | 4 (5)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Body aches (General disorders) | 1 (1) | 0 (0) | 0 (0)
Finger and cuticle pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Myocardial bridge, murmur (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Eye redness (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Elevated Carcinoembryonic Antigen (Investigations) | 0 (0) | 0 (0) | 3 (3)
Torn Left Rotator Cuff (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle spasm (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Narcotic withdrawal (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Restless legs (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Benign prostate hyperplasia (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Adenocarcinoma of transverse colon (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Left arm pit rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Back spasm (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Weight loss (Investigations) | 1 (2) | 2 (2) | 5 (5)
Weight gain (Investigations) | 0 (0) | 1 (1) | 0 (0)
watering eyes (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
white blood cell decreased (Investigations) | 1 (2) | 4 (12) | 2 (4)
Platelet count decreased (Investigations) | 1 (1) | 1 (1) | 3 (4)
Cholesterol high (Investigations) | 0 (0) | 0 (0) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (3) | 1 (1) | 8 (9)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (4)
Rash acneiform (Skin and subcutaneous tissue disorders) | 3 (4) | 7 (10) | 11 (17)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4) | 4 (4)
Hypertrichosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 2 (2) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 2 (2)
Small intestinal mucositis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Mucosal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 2 (2)
History of Medullary Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 11 (11)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (3)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Skin on eye lids irritated (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Nail loss (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 2 (2) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-06): https://cdn.clinicaltrials.gov/large-docs/29/NCT03263429/Prot_SAP_001.pdf
  • Informed Consent Form (2022-01-18): https://cdn.clinicaltrials.gov/large-docs/29/NCT03263429/ICF_000.pdf